CLINICAL TRIAL: NCT07100561
Title: Extensive Post-discharge Counselling and Phone-based Follow-up Intervention to Reduce Heart Failure Readmission- A Pilot Randomized Control Trial
Brief Title: 30 Days and 90 Days Heart Failure Re-Admission at Komfo Anokye Teaching Hospital
Acronym: HeFRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Komfo Anokye Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KATHIRB/AP/031/25
Record Dates: First submitted 2025-07-01; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: heart failure readmission; phone-based follow up; extensive post discharge counseling; pilot randomized control trial
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control/Usual Care (No Intervention): The usual care (counselling by their attending physicians and their normal outpatient reviews).
- intervention arm (Experimental)
  Interventions: Other: Extensive post discharge counselling and phone-based follow up

INTERVENTIONS:
Other: Extensive post discharge counselling and phone-based follow up — Counselling by their attending physicians plus Extensive post-discharge counselling from a study doctor/pharmacist/a trained nurse and telephone follow-ups in addition to their normal outpatient reviews. The telephone follow-ups will be weekly for the first 30 days and then 4 weekly till day 90.
  Arms: intervention arm

SUMMARY:
In Ghana, about 88.3 per cent of cardiac admissions are due to Heart failure, making it the leading cause of admission due to heart conditions. Despite improved knowledge on heart failure and an increasing array of evidence-based guideline treatment options, there is still a significant readmission rate worldwide. This may be due to the underutilization of these evidence-based therapies or a lack of proper follow-up on these patients. Recurrent hospital admission is an independent predictor of death in heart failure. Strategies aimed at providing increased support at discharge and effective follow-up may be associated with lower readmission risk. This study aims to assess the effect of extensive post-discharge counselling and effective phone-based follow-up on the 30-day and 90-day heart failure readmission rate at a tertiary hospital in Ghana. This is a single-centre, pilot randomised controlled trial of heart failure patients admitted to the Komfo Anokye Teaching Hospital

ELIGIBILITY:
Inclusion Criteria:

* · Adults Aged 18 years and above

  * Diagnosed with heart failure
  * NYHA Class II-IV
  * Informed consent

Exclusion Criteria:

* · NHYA class I

  * Patients who do not have access to a mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
30-day and 90-day heart failure readmissions between the intervention group and the control group. | 90 days
  30-day and 90-day heart failure readmissions between the intervention group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ashanti Region, Ghana

IPD SHARING:
Plan to Share IPD: Undecided